CLINICAL TRIAL: NCT02749669
Title: Health Care Courses of Elderly Hospitalized Patients for Inappropriate Reasons: Qualitative and Economic Analyzes
Acronym: PAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Régis AUBRY (Other)
Responsible Party: Sponsor-Investigator, Régis AUBRY, Professor, Centre Hospitalier Universitaire de Besancon
Organization: Centre Hospitalier Universitaire de Besancon (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAGE
Record Dates: First submitted 2016-04-07; First posted 2016-04-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-04

CONDITIONS: Cognitive Impairment
Keywords: Inappropriate hospitalization; elderly; mild or moderate cognitive impairment; qualitative research; economic evaluation
MeSH Terms: conditions — Cognitive Dysfunction; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qualitative research (Other): Semi-structured interviews
  Interventions: Other: Qualitative research
- Economic evaluation (No Intervention): Questionnaire

INTERVENTIONS:
Other: Qualitative research — Semi-structured Interviews
  Arms: Qualitative research

SUMMARY:
For almost 17 % of cases patients over 75 years are sent for inappropriate reasons to the emergency unit. They are described as inappropriate hospitalization because they don't require the use of technical platform or diagnostic neither therapeutic procedures under medical supervision. Those are inappropriate because the patient could have a paramedical and social care at home or in more efficient structures. The hospital remains the place of remedy for social and health situations whose resolution was not possible because of a lack of infrastructure available, of patient or his relative information, or a lack of coordination in medico-social establishment.

These inappropriate hospitalizations involve an increase of length of stay that enhancing the fragility and vulnerability of the elderly. They have deleterious effects as decompensation, comorbidities and loss of autonomy.

Moreover, the suffering of natural or informal caregivers is also an important public health question; Caregivers may have a serious disease resulting from caring their relative. That leads to increase their consumption of health care and medical goods.

This comprehensive study will highlight the deficiencies of the actual health care through the analysis of the speech of the different parts involved (main study). Simultaneously, a comparative analysis of the costs of health care will be conducted (economic combined study).

DETAILED DESCRIPTION:
For almost 17 % of cases patients over 75 years are sent for inappropriate reasons to the emergency unit. They are described as inappropriate hospitalization because they don't require the use of technical platform or diagnostic neither therapeutic procedures under medical supervision. Those are inappropriate because the patient could have a paramedical and social care at home or in more efficient structures. The hospital remains the place of remedy for social and health situations whose resolution was not possible because of a lack of infrastructure available, of patient or his relative information, or a lack of coordination in medico-social establishment.

These inappropriate hospitalizations involve an increase of length of stay that enhancing the fragility and vulnerability of the elderly. They have deleterious effects as decompensation, comorbidities and loss of autonomy.

Moreover, the suffering of natural or informal caregivers is also an important public health question; Caregivers may have a serious disease resulting from caring their relative. That leads to increase their consumption of health care and medical goods.

This comprehensive study will highlight the deficiencies of the actual health care through the analysis of the speech of the different parts involved (main study). Simultaneously, a comparative analysis of the costs of health care will be conducted (economic combined study).

When a patient over 75 years will arrive in the emergency or geriatrics units of the University Hospital of Besançon and the reason for admission indicated in the hospital record will be " difficult home care " or " caregiver burn out " or any other reason unjustified from a strictly medical point of view, the investigator will ensure the patient's eligibility under the inclusion and non-inclusion criteria, and will do a review of appropriateness of hospital according Appropriate Assessment Protocol criteria.

All patients corresponding to the inclusion criteria during the three months of the inclusion period will be identified in the reference population. Expected active file is fifteen patients in three months. The reference population of patients in the active file will be followed for six months. Steps of their health care will be identified and described in a questionnaire detailing the patient's pathway by collecting data on:

* Dates when they change their place of living or care,
* Places of living or care at every step.

The qualitative study will include five patients of the reference population in order to describe, analyze and understand in depth their health care through semi-structured interviews. To analyze a variety of pathways, 5 patients will be selected in order to represent the heterogeneity of admission places (emergency or geriatric unit), as well as the places of origin (home institution).

The interview will be also proposed to relevant people involved (health professionals, professional home) in the situation and at least to one relative designated by the patient.

For each change of place of residence or place of care (or return at home) of the five patients, the interviews will be conducted with the patient and relevant stakeholders.

At the end of the first step, the investigator will join to the outgoing mail, a document to ensure that the later steps of patient health care is collected. For each step, the referring health professional will have to do the same in order to compile data of the patient's pathway.

Thus, from an estimate of three key steps to describe and analyze the healthcare trajectories of five patients during six months, 90 interviews will be conducted, transcribed and analyzed.

The economic combined study will focus on the five patients followed in the qualitative study. This descriptive and prospective study will analyze the differential costs between the actual health care course and a more appropriate care course. The study will be conducted according to a "societal" perspective.

The most appropriate health care courses will be selected by healthcare professionals who specialize in elderly care in the Besançon area (medical structures, gerontological network…). The patients actual care courses will be presented to them and they will collectively decide which care course would have been most appropriate for each patient.

The costs of the actual and most appropriate courses will be evaluated as follows:

* Direct medical costs regarding hospitalizations, consultations, medical and technical procedures, laboratory and pathology costs, and medical transport expenses.
* Direct non-medical costs regarding social expenses (accommodation). Welfare received by the elderly patients; expenses of the elderly patients or their relatives related to special facilities and adaptation of the home. Allowances received by relatives in case of sick leave and the cost associated with consumption of medication and medical transport (sleep disorders, anxiety and depression, nutritional and memory disorders, cardiovascular disorders including hypertension, decompensation of chronic diseases...).

These costs will be collected:

* in the patient's medical record,
* in the record compiled by the social worker,
* in the databases of Regional Health Authority of Franche-Comté
* in the hospital Discharge Abstract Database (PMSI)
* as well as with a questionnaire to patients and caregivers.

The global expenditure related to the actual care course and the most appropriate course as defined by healthcare professionals will be calculated.

Finally, this economic combined study will analyze the differential costs between current patient health care and a more relevant patient health care.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years old and older,
* Hospitalized in the emergency or geriatric units of the University Hospital of Besançon for inappropriate reasons according to Appropriate Assessment Protocol criteria,
* With a history of mild to moderate cognitive impairment according to the latest cognitive assessment (HAS 2009),
* Who have expressed no objection towards collecting and processing personal data (health care, health status, demographic and socio-economic characteristics) after information regarding the goals and course of the study.
* Adults under guardianship may be included

For the five patients followed:

* Able to speak French,
* Who have given their written consent to participate in the study after information about the objectives and course of the study (interviews, collection of personal data).

Exclusion Criteria:

- Patients who have expressed their opposition to collecting and processing personal data.

For the five patients followed:

* Patients with a history of cognitive impairment preventing the semi-structured interview,
* Unable to speak French.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
90 semi-structured interviews | 6 months
  Qualitative Data analysis - Theoretical saturation

SECONDARY OUTCOMES:
Demographic and socio-economic questionnaires of 15 patients | 6 months
  Socio-economic analysis
Caregiver Reaction Assessment (CRA) scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Séverine KOEBERLE, Dr, Principal Investigator — Centre Hospitalier Universitaire de Besancon; Thomas TANNOU, Dr, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- AUBRY Regis, Besançon, France